CLINICAL TRIAL: NCT05976464
Title: Efficacy of Magnesium Sulfate as an Adjuvant to Local Anesthetic in Erector Spinae Plane Block for Post-operative Analgesia After Modified Radical Mastectomy
Brief Title: Efficacy of Magnesium Sulfate as an Adjuvant in Erector Spinae Plane Block as an Anesthetic Post Operative After Modified Radical Mastectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doha Mohamed Ahmed, MD, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: magnesium analgesic efficacy
Record Dates: First submitted 2023-07-13; First posted 2023-08-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: ESPB, Mg Sulfate,Post Mastectomy
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium sulphate as an adjuvant to local anesthetic in erector spinae plane block (Active Comparator): Ultrasound-guided Erector spinae plane (ESP) block will be done with the patient in a sitting position depending on the surgical site (lt. or Rt.) ESP block will be given using high-frequency linear u/s transducer, the probe is placed in longitudinal orientation lateral to the thoracic third and sixth spinous process, the erector spinae muscle, is identified from the surface, we will deposit 20 ml of 0.25% levobupivacaine into interfacial plane below erector spinae muscle.
  Interventions: Drug: Magnesium sulfate in erector spinae plane block
- local anesthetic only in erector spinae plane block (Experimental): Ultrasound-guided Erector spinae plane (ESP) block will be done with the patient in a sitting position depending on surgical site (lt. or Rt.) ESP block will be given using high-frequency linear u/s transducer, the probe is placed in longitudinal orientation lateral to the thoracic third and sixth spinous process, the erector spinae muscle, is identified from the surface, we will deposit 20 ml of 0.25% levobupivacaine and magnesium sulfate into interfacial plane below erector spinae muscle.
  Interventions: Drug: Magnesium sulfate in erector spinae plane block

INTERVENTIONS:
Drug: Magnesium sulfate in erector spinae plane block — Ultrasound-guided Erector spinae plane (ESP) block will be done with the patient in a sitting position depending on the surgical site (lt. or Rt.) ESP block will be given using high-frequency linear u/s transducer, the probe is placed in longitudinal orientation lateral to the thoracic third and sixth spinous process, the erector spinae muscle, is identified from the surface, we will deposit 20 ml of 0.25% levobupivacaine into interfacial plane below erector spinae muscle.
  General anesthesia will be induced with l/kg fentanyl, 2mg/kg propofol, 0.5 mg/kg atracurium and inhalational anesthesia (sevoflurane) No other narcotic, analgesic or sedative will be administrated during the operative period.
  BP(SystolicBP, DiastolicBP) and HR will be observed and recorded every 30 min till the end of surgery.

SUMMARY:
efficacy of magnesium sulfate as an adjuvant in erector spinae plane block as an anesthetic post-operative after modified radical mastectomy

DETAILED DESCRIPTION:
magnesium sulphate as an adjuvant to local anesthetic in erector spinae plane block compared to local anesthetic only in erector spinae plane block

ELIGIBILITY:
Inclusion Criteria:

* 1. ASA I-II. 2. Female patients aged 18-65 years. 3. Scheduled for a modified radical mastectomy with axillary dissection for breast cancer.

Exclusion Criteria:

1. ASA < II.
2. more than 65 years old
3. Patients with known allergies to the study drugs
4. Skin infection at the site of needle puncture.
5. Coagulopathy

5. Drug or as that would interfere with perception and assessment of pain. 6. Uncooperative patients.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
- The primary outcome measure in this study will be the total dose of morphine consumption during the 24 hour Postoperatively. | Up to 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: mohamed a.m bakr, professor, Study Chair — professor of anesthesia
Locations (1):
- Assuit University -South Egypt Cancer Institute, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No